CLINICAL TRIAL: NCT06948357
Title: A Multicenter, Randomized, Double-Blind, Crossover, Placebo-Controlled Phase II Clinical Study to Evaluate the Efficacy and Safety of BRIMOCHOL PF, CARBACHOL PF in Chinese Patients With Presbyopia
Brief Title: Efficacy and Safety of BRIMOCHOL PF and CARBACHOL PF in Chinese Presbyopia Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhaoke (Guangzhou) Ophthalmology Pharmaceutical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZKO-CSP-BRI-CAR-201
Record Dates: First submitted 2025-03-06; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-02

CONDITIONS: Presbyopia
Keywords: presbyopia; eye drops; ophthalmic solution; Chinese; Brimochol; Carbachol; Brimonidine
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Treatment Sequences 1 (Experimental): BRIMOCHOL PF eye drops and placebo eye drops given once respectively in visit 2; CARBACHOL PF eye drops and placebo eye drops given once respectively in visit 3; Brimonidine eye drops and placebo eye drops given once respectively in visit 4; BRIMOCHOL PF eye drops given twice in visit 5; CARBACHOL PF eye drops given twice in visit 6; Brimonidine eye drops given twice in visit 7; Placebo eye drops given twice in visit 8.
  Interventions: Drug: BRIMOCHOL PF eye drops; CARBACHOL PF eye drops; Brimonidine eye drops; Placebo
- Treatment Sequences 2 (Experimental): Placebo eye drops given twice in visit 2; BRIMOCHOL PF eye drops and placebo eye drops given once respectively in visit 3; CARBACHOL PF eye drops and placebo eye drops given once respectively in visit 4; Brimonidine eye drops and placebo eye drops given once respectively in visit 5; BRIMOCHOL PF eye drops given twice in visit 6; CARBACHOL PF eye drops given twice in visit 7; Brimonidine eye drops given twice in visit8.
  Interventions: Drug: BRIMOCHOL PF eye drops; CARBACHOL PF eye drops; Brimonidine eye drops; Placebo
- Treatment Sequences 3 (Experimental): Brimonidine eye drops given twice in visit 2; Placebo eye drops given twice in visit 3; BRIMOCHOL PF eye drops and placebo eye drops given once respectively in visit 4; CARBACHOL PF eye drops and placebo eye drops given once respectively in visit 5; Brimonidine eye drops and placebo eye drops given once respectively in visit 6; BRIMOCHOL PF eye drops given twice in visit 7; CARBACHOL PF eye drops given twice in visit 8.
  Interventions: Drug: BRIMOCHOL PF eye drops; CARBACHOL PF eye drops; Brimonidine eye drops; Placebo
- Treatment Sequences 4 (Experimental): CARBACHOL PF eye drops given twice in visit 2; Brimonidine eye drops given twice in visit 3; Placebo eye drops given twice in visit 4; BRIMOCHOL PF eye drops and placebo eye drops given once respectively in visit 5; CARBACHOL PF eye drops and placebo eye drops given once respectively in visit 6; Brimonidine eye drops and placebo eye drops given once respectively in visit 7; BRIMOCHOL PF eye drops given twice in visit 8.
  Interventions: Drug: BRIMOCHOL PF eye drops; CARBACHOL PF eye drops; Brimonidine eye drops; Placebo
- Treatment Sequences 5 (Experimental): BRIMOCHOL PF eye drops given twice in visit 2; CARBACHOL PF eye drops given twice in visit 3; Brimonidine eye drops given twice in visit 4; Placebo eye drops given twice in visit 5; BRIMOCHOL PF eye drops and placebo eye drops given once respectively in visit 6; CARBACHOL PF eye drops and placebo eye drops given once respectively in visit 7; Brimonidine eye drops and placebo eye drops given once respectively in visit 8.
  Interventions: Drug: BRIMOCHOL PF eye drops; CARBACHOL PF eye drops; Brimonidine eye drops; Placebo
- Treatment Sequences 6 (Experimental): Brimonidine eye drops and placebo eye drops given once respectively in visit 2; BRIMOCHOL PF eye drops given twice in visit 3; CARBACHOL PF eye drops given twice in visit 4; Brimonidine eye drops given twice in visit 5; Placebo eye drops given twice in visit 6; BRIMOCHOL PF eye drops and placebo eye drops given once respectively in visit 7; CARBACHOL PF eye drops and placebo eye drops given once respectively in visit 8.
  Interventions: Drug: BRIMOCHOL PF eye drops; CARBACHOL PF eye drops; Brimonidine eye drops; Placebo
- Treatment Sequences 7 (Experimental): CARBACHOL PF eye drops and placebo eye drops given once respectively in visit 2; Brimonidine eye drops and placebo eye drops given once respectively in visit 3; BRIMOCHOL PF eye drops given twice in visit 4; CARBACHOL PF eye drops given twice in visit 5; Brimonidine eye drops given twice in visit 6; Placebo eye drops given twice in visit 7; BRIMOCHOL PF eye drops and placebo eye drops given once respectively in visit 8.
  Interventions: Drug: BRIMOCHOL PF eye drops; CARBACHOL PF eye drops; Brimonidine eye drops; Placebo

INTERVENTIONS:
Drug: BRIMOCHOL PF eye drops; CARBACHOL PF eye drops; Brimonidine eye drops; Placebo — BRIMOCHOL PF eye drops, CARBACHOL PF eye drops, Brimonidine eye drops and Placebo were administered in 7 treatment sequences in various combinations and doses

SUMMARY:
A multicenter, randomized, double-Blind, crossover, placebo-controlled Phase II clinical Study to evaluate the efficacy and safety of BRIMOCHOL PF and CARBACHOL PF in the treatment of Chinese patients with presbyopia.

DETAILED DESCRIPTION:
119 subjects were planned to be enrolled in this study and randomly assigned in equal proportions into 7 treatment sequences. Each subject will receive a total of 7 treatments, each treatment period will be 1 day, and two adjacent visits during the treatment period need to be eluted for at least 3 days。

The study period included the screening period (Day 14~Day 1) with 1 visit and the treatment period (Day 0~Day 30) with 7 visits. There were a total of 8 visits in this study, with a duration of 32 to 45 days.

ELIGIBILITY:
Inclusion Criteria:

1. At Visit 1 (Screening Period), the age ranges from 45 to 75 years old, regardless of gender
2. At Visit 1 (Screening Period), the corrected distance visual acuity of either eye is ≥ 0.8 (National Standard Logarithmic Visual Acuity Scale,decimal visual acuity) in the clinical routine manifest refraction (distance vision).
3. At Visit 1 (Screening Period), the manifest refraction (distance vision under mesopic conditions) results are as follows: For any eye,-4.00D ≤ equivalent spherical lens power ≤ +2.00D, and the negative cylinder lens power is ≥-2.00D;
4. At least one eye meeting the following at both Visit 1 and Visit 2:

   1. Under mesopic conditions, monocular corrected near visual acuity (MCNVA) ≤65 ETDRS letters (equivalent to decimal visual acuity 0.4) ;
   2. Under mesopic conditions, monocular corrected near visual acuity with a multiple-pinhole occluder (MCNVA_P) improves by ≥15 ETDRS letters compared to monocular corrected near visual acuity without the occluder (MCNVA).
5. During Visit 1 (Screening Period) and Visit 2, both eyes must meet the following criteria:under mesopic conditions, binocular corrected near visual acuity (BCNVA) is ≤65 ETDRS letters (equivalent to decimal visual acuity 0.4);
6. Any eye is phakic or implanted with a monofocal intraocular lens (IOL);
7. Normal iris and pupillary morphology in any eye, with normal light reflex and an interocular pupillary diameter difference ≤1 mm during screening;

Exclusion Criteria:

1. Use of corneal or scleral contact lenses within 28 days prior to screening or planned for the duration of the study;
2. Narrow anterior chamber angle (Van Herick grade ≤2 via slit lamp examination) or previous iridotomy or resection in either eye；
3. Ocular history in any eye: hyphema, ciliary body detachment, iridodonesis, or ocular trauma；
4. Any eye with a corneal abnormality that, in the judgment of the investigator, affects visual acuity or intraocular pressure measurements, including moderate to severe dry eye (e.g., significant signs of ocular surface damage (≥5 corneal fluorescein staining spots) on slit lamp microscopy);
5. Any phakic eye has a history of lens tremor, subluxation, or suspected zonular laxity; or any pseudophakic eye has undergone posterior capsulotomy or uses multifocal or extended depth of focus intraocular lenses.
6. Any eye with an axial length of ≥26mm;
7. Either eye has undergone intraocular or corneal surgery (only non-complicated cataract surgery with a monofocal lens placed in the capsular bag more than 6 months after the date of surgery is permitted; complicated cataract surgery is defined as surgery that has resulted in a rupture of the capsule or placement of an IOL outside the capsule (ciliary sulcus, scleral or iris fixation, anterior chamber, etc.));
8. Either eye has a history of congenital or traumatic cataract, congenital aphakia, or opacities in the refractive media that affect visual acuity in the visual axis area.
9. History of uveitis, low intraocular pressure (IOP < 9 mmHg), glaucoma or hypertension (IOP > 21 mmHg) or pseudoexfoliation syndrome in either eye;
10. Active ocular or periocular infection or inflammation in either eye, or a history of recurrent infection or chronic infection (e.g., herpes virus infection) in either eye;
11. Either eye has a history of retinal diseases (such as retinal detachment, age-related macular degeneration, diabetic retinopathy, peripheral retinal diseases that increase the risk of the subject as judged by the investigator) or optic nerve abnormalities.
12. During the screening period, any eye has any ocular disease other than presbyopia that requires treatment with ocular preparations, intravitreal injection or ocular surgery during the study period (except artificial tears, which can be used on the day of ocular examination during the screening period and on non-treatment visits).

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Estimated)
Dates: Start 2025-03-24 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes in MCNVA(monocular corrected near visual acuity) ETDRS letters and MCDVA (monocular corrected distance visual acuity) ETDRS letters from baseline in the study eyes after administration | 15minutes, 1hour, 2hour, 4hour15minutes, 6hour, and 8hour after administration
  In the mesopic condition, the proportion of subjects whose MCNVA in the study eye increased by ≥15 ETDRS letters and whose MCDVA in the study eye did not decrease by ≥5 ETDRS letters from the pre-dose baseline at 15minutes, 1hour, 2hour, 4hour15minutes, 6hour, and 8hour after dosing.

SECONDARY OUTCOMES:
Changes in MCNVA(monocular corrected near visual acuity) ETDRS letters from baseline in the study eyes after administration | 15minutes, 1hour, 2hour, 4hour15minutes, 6hour, and 8hour after administration
  1. In the mesopic conditions, the proportion of subjects whose MCNVA in the study eye increased by ≥ 10 ETDRS letters and whose MCDVA in the study eye did not decrease by ≥5 ETDRS letters from the pre-dose baseline at 15minutes, 1hour, 2hour, 4hour15minutes, 6hour, and 8hour after dosing.
  2. In the mesopic conditions, the proportion of subjects whose MCNVA in the study eye increased by ≥ 15 ETDRS letters from the pre-dose baseline at 15minutes, 1hour, 2hour, 4hour15minutes, 6hour, and 8hour after dosing.
  3. In the mesopic conditions, the proportion of subjects whose MCNVA in the study eye increased by ≥ 10 ETDRS letters from the pre-dose baseline at 15minutes, 1hour, 2hour, 4hour15minutes, 6hour, and 8hour after dosing.
Changes in MCNVA(monocular corrected near visual acuity) ETDRS letters from baseline in the study eyes after administration | 15 minutes to 8 hours after administration
  Mean ETDRS letter gain in study eye MCNVA compared to the baseline measurements under mesopic conditions across all post-dose evaluation intervals (15 minutes through 8 hours).
Changes in MCNVA(monocular corrected near visual acuity) ETDRS letters from baseline in the study eyes after administration | 15 minutes to 8 hours after administration
  The weighted mean of the area under the curve (AUC) for the increase in MCNVA ETDRS letter gain from baseline under mesopic conditions in the study eye across post-dose evaluation intervals (15 minutes through 8 hours).
Changes in BCNVA (Binocular Corrected Near Visual Acuity) ETDRS letters and BCDVA (Binocular Corrected Distance Visual Acuity) ETDRS letters from baseline after administration | 15minutes, 1hour, 2hour, 4hour15minutes, 6hour, and 8hour after administration
  1. In the mesopic condition, the proportion of subjects whose BCNVA increased by ≥15 ETDRS letters and whose BCDVA did not decrease by ≥5 ETDRS letters from the pre-dose baseline at 15minutes, 1hour, 2hour, 4hour15minutes, 6hour, and 8hour after dosing.
  2. In the mesopic condition, the proportion of subjects whose BCNVA increased by ≥10 ETDRS letters and whose BCDVA did not decrease by ≥5 ETDRS letters from the pre-dose baseline at 15minutes, 1hour, 2hour, 4hour15minutes, 6hour, and 8hour after dosing.
  3. In the mesopic conditions, the proportion of subjects whose BCNVA increased by ≥ 15 ETDRS letters across all post-dose evaluation intervals (15minutes through 8hour).
  4. In the mesopic conditions, the proportion of subjects whose BCNVA increased by ≥ 10 ETDRS letters across all post-dose evaluation intervals (15minutes through 8hour).
Changes in pupil diameter from baseline after administration | 15minutes, 1hour, 2hour, 4hour15minutes, 6hour, and 8hour after administration
  Quantitative changes in pupil diameter (measured in study eye and binocular average) from pre-dose baseline values under mesopic conditions at 15minutes, 1hour, 2hour, 4hour15minutes, 6hour, and 8hour after administration.

CONTACTS AND LOCATIONS:
Overall Officials: Jia Qu, Principal Investigator — Optometry Hospital of Wenzhou Medical University
Locations (1):
- Optometry Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No